CLINICAL TRIAL: NCT03186144
Title: Clinical and Molecular Study of CHARGE Syndrom
Acronym: CHARGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Diagnostic
Other Study IDs: CHARGE
Record Dates: First submitted 2016-08-26; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Development Abnormalies; Inclusion on Clinical Criteria of the Syndrome
MeSH Terms: interventions — Genetic Testing

ARMS (1):
- No arm : descriptive study (Experimental)
  Interventions: Genetic: Blodd punction for genetic analysis

INTERVENTIONS:
Genetic: Blodd punction for genetic analysis

SUMMARY:
1. Clinical description of a French cohort of patients with CHARGE syndrome.
2. Search any phenotype-genotype correlation in typical, atypical or incomplete form of the syndrome
3. Using Next generation Sequencing, try to identify other genes involved in this syndrome, as the CHD7 gene is involved in only 40-60% of cases

ELIGIBILITY:
Inclusion Criteria: Clinical criteria

Major criteria:

* Ocular coloboma
* Chonamal atresia and/or cleft palate
* Semi-CircularCanals hypoplasia

Minor criteria:

* Cranial nerves
* Hypothalamic-pituitary deficiency
* Internal or external ear malformation
* Cardiac, esophageal malformations
* Intellectual Deficiency

Diagnosis criteria:

* Typical CHARGE: 3 major criteria or 2 major + 2 minor
* Partial CHARGE: 2 major + 1 minor
* Atypical CHARGE: 2 major without minor or 1 major + 2 minor

Exclusion Criteria:

* Absent consentment for genetic analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Description Clinical and molecular analysis of a French cohort CHARGE | 12 month
Execution of the socio-adaptive scale, parental scale | 12 month
Rate of mutations of CHD7 and / or type of mutations | 12 month
analysis CHD7 gene from the patient's DNA | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- French Referent centers for developement abnomalies, Poitiers, France